CLINICAL TRIAL: NCT05963139
Title: Comparison of Local Anesthetic Dose in IPACK (Interspace Between the Popliteal Artery and the Posterior Capsule of the Knee) Block Performed for Postoperative Analgesia in Knee Artroplasty Operations
Brief Title: Comparison of Local Anesthetic Dose in Ipack Block Performed in Knee Arthroplasty Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-1481345
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Analgesia; Pain, Postoperative; Anesthesia
Keywords: IPACK block; Postoperative Pain; Postoperative Patient Controlled Analgesia; Knee Artroplasty; Regional Anesthesia; Numeric rating scale
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1:10 ml %0,25 bupivacaine ıpack and 15 ml %0,25 bupivacaine adductor block (Active Comparator): In this group,US guided IPACK block will be performed with 10 ml %0,25 bupivacaine and adductor block will be performed with 15 ml %0.25 bupivacaine using a 22 gauge 10 mm block needle.
  Interventions: Drug: Bupivacaine; Drug: Morphine Sulfate
- Group 2:15 ml %0,25 bupivacaine ıpack and 15 ml %0,25 bupivacaine adductor block (Active Comparator): In this group,US guided IPACK block will be performed with 15 ml %0,25 bupivacaine and adductor block will be performed with 15 ml %0.25 bupivacaine using a 22 gauge 10 mm block needle.
  Interventions: Drug: Bupivacaine; Drug: Morphine Sulfate
- Group 3:20 ml %0,25 bupivacaine ıpack and 15 ml %0,25 bupivacaine adductor block (Active Comparator): In this group,US guided IPACK block will be performed with 20 ml %0,25 bupivacaine and adductor block will be performed with 15 ml %0.25 bupivacaine using a 22 gauge 10 mm block needle.
  Interventions: Drug: Bupivacaine; Drug: Morphine Sulfate
- Group 4:15 ml %0,25 bupivacaine adductor block and intravenous patient controlled analgesia (Active Comparator): In this group adductor block will be performed with 15 ml %0.25 bupivacaine using a 22 gauge 10 mm block needle and postoperative patient controlled analgesia with morphine will be preferred for postoperative analgesia method.
  Interventions: Drug: Bupivacaine; Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Bupivacaine — US guided IPACK block will be performed with 10/15/20 ml %0,25 bupivacaine and adductor block will be performed with 15 ml %0,25 bupivacaine.
  Other Names: Marcaine
Drug: Morphine Sulfate — In this group,adductor block will be performed with 15 ml %0,25 bupivacaine using a 22 gauge 10 mm block needle and patients will be postoperatively administered patient controlled analgesia with morphine.
  Other Names: morphine

SUMMARY:
The investigators research was designed as a single-center, prospective, randomized study. The patients undergoing knee artrhroplasty surgery in Istanbul University Istanbul Medicine Faculty Department of Orthopedics and Traumatology will be included. Patients who are legally authorized to make decisions on their behalf will be informed about the research and their written consent will be obtained. Patients who do not give consent will not be included in the study.

Patients will be given US guided IPACK and adductor blocks using a 22 gauge 10 mm block needle after compliance with the rules of asepsia and antisepsis in the supine position according to the group of patients in which they were included.

IPACK and adductor block will be done for postoperative analgesia. After then, a single dose of spinal anesthesia will be applied as a regional anesthesia method, in a sitting position, using the appropriate spinal needle, as is routinely applied in the investigators clinic. After the block is completed, the pinprick test will be done and the operation will be started after the successful completion of the block is confirmed. Oxygen will be given to the patients with a face mask at 4 lt / min throughout the operation. ECG, saturation, invasive / noninvasive blood pressure monitoring of the patients will be done.

In the investigators clinic, the use of IPACK block, adductor block and PCA (patient controlled analgesia) device with intravenous morphine for postoperative analgesia is routinely performed. In this study, four randomized groups will be formed together with the control group.

IPACK block will be applied to the 1st group with 10 ml of 0.25% bupivacaine, to the 2nd group with 15 ml of 0.25% bupivacaine, and to the 3rd group with 20 ml of 0.25% bupivacaine.Adductor block will be applied to all the groups with 15 ml %0,25 bupivacaine and PCA (patient controlled analgesia) device with intravenous morphine for postoperative analgesia is performed.

Pain score and total morphine consumption will be determined by numeric rating scale (NRS) at the postoperative 1, 4, 8, 12, 24 and 48th hours by providing the use of a PCA device with intravenous morphine applied in routine practice to all four groups. As in routine practice, when NRS > 4 after each interrogation, morphine 2 mg iv will be administered as additional analgesia and the maximum will be increased to 10 mg. Pain management will continue when NRS < 4.

DETAILED DESCRIPTION:
The investigators research was designed as a single-center, prospective, randomized study.

The patients undergoing knee arthroplasty in Istanbul University Istanbul Medicine Faculty Department of Orthopedics and Traumatology will be included. Patients who are legally authorized to make decisions on their behalf will be informed about the research and their written consent will be obtained. Patients who do not give consent will not be included in the study.

Patients will be evaluated preoperative before surgery, a detailed history will be taken and physical examination will be carried out. Medical and surgical resume information will be obtained. Patients' NRS scores will be recorded before the operation. Patients will be taken to the operating room after premedication.

ECG, pulse oximeter, blood pressure monitoring will be performed in the operating room. Patients will be given US guided IPACK and adductor blocks using a 22 gauge 10 mm block needle after compliance with the rules of asepsia and antisepsis in the supine position according to the group of patients in which they were included.

IPACK and adductor block will be done for postoperative analgesia. After then, a single dose of spinal anesthesia will be applied as a regional anesthesia method, in a sitting position, using the appropriate spinal needle, as is routinely applied in the investigators clinic. After the block is completed, the pinprick test will be done and the operation will be started after the successful completion of the block is confirmed. Oxygen will be given to the patients with a face mask at 4 lt / min throughout the operation.ECG, saturation, invasive / noninvasive blood pressure monitoring of the patients will be done.

In the investigators clinic, the use of IPACK block, adductor block and PCA (patient controlled analgesia) device with intravenous morphine for postoperative analgesia is routinely performed. In this study, four randomized groups will be formed together with the control group.Computer-generated random numbers will be used for simple randomization of patients.

IPACK block will be applied to the 1st group with 10 ml of 0.25% bupivacaine, to the 2nd group with 15 ml of 0.25% bupivacaine, and to the 3rd group with 20 ml of 0.25% bupivacaine.Adductor block will be applied to all the groups with 15 ml %0,25 bupivacaine and PCA (patient controlled analgesia) device with intravenous morphine for postoperative analgesia is performed.

Pain score and total morphine consumption will be determined by numeric rating scale (NRS) at the postoperative 1, 4, 8, 12, 24 and 48th hours by providing the use of a PCA device with intravenous morphine applied in routine practice to all four groups. As in routine practice, when NRS > 4 after each interrogation, morphine 2 mg iv will be administered as additional analgesia and the maximum will be increased to 10 mg. Pain management will continue when NRS < 4.

Patients are followed up in the service for 48 hours postoperatively in routine practice.

In the postoperative period, patients will be evaluated in terms of additional nausea and vomiting,amount of morphine consumed and additional analgesic need postoperative period up to 48 hours.First mobilization time, hospitalization time will be evaluated.Womac osteoarthritis index and joint range of motion will be evaluated at preoperative period and at the discharge day from the hospital.The Medical Research Council (MRC) Scale for Muscle Strength for lower extremity will be evaluated preoperative period, at postoperative 24th hour and at the discharge day from the hospital.

Postop patient satisfaction and surgical satisfaction with Likert scale will also be evaluated at postoperative period.

During the procedure, complications such as failed block, nerve damage, vascular injury, intravenous injection of local anesthetic, local anesthetic toxicity and allergic reactions will be recorded.

Before the study, it was determined that at least 112 patients should be collected in the power analysis performed with the help of similar literature data. After collecting the demographic data and morphine consumption data of the patients, the data will be transferred to the statistical program called SPSS and statistical analysis will be made.The investigators study does not contain any modifications other than the investigators daily routine practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for knee arthroplasty surgery under regional anesthesia
* ASA(American Society of Anesthesiology) 1-3
* Receiving consent that accept regional analgesia

Exclusion Criteria:

* Refusal of regional anesthesia
* Infection on the local anesthetic application area
* Infection in the central nervous system
* Coagulopathy
* BMI > 40
* Known allergy against local anesthetics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(0-10)pain scores for patients. | postoperative period up to 48 hours
  NRS(Numeric Rating Scale),0:no pain,10:the worst pain.
Opioid (mg) consumption | postoperative period up to 48th hours
  Opioid (mg) consumption

SECONDARY OUTCOMES:
Incidence of side effects | postoperative period up to 48th hours
  Incidence of nausea and vomiting
Time until postoperative first mobilization | Up to 48 hours
  First mobilization time
Length of hospital stay | Through study completion, an average of 1 week.
  Hospitalization
Womac osteoarthritis index | Discharge 1 day from the hospital
  Womac osteoarthritis index
The Medical Research Council (MRC) Scale for Muscle Strength for lower extremity | Discharge 1 day from the hospital
  The Medical Research Council (MRC) Scale for Muscle Strength is a commonly used scale for assessing muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction).
Joint range of motion | Postoperative period up to 48th hours, discharge 1 day
  Joint range of motion
Patient satisfaction | Postoperative period up to 48th hours
  Satisfaction score;0-very unsatisfied,5-very satisfied.
Surgeon satisfaction | Postoperative period up to 48th hours
  Satisfaction score;0-very unsatisfied,5-very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLBERK KILIÇ, MD, Principal Investigator — Istanbul Faculty of Medicine
Locations (1):
- Istanbul University Istanbul Medical Faculty, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Zheng FY, Liu YB, Huang H, Xu S, Ma XJ, Liu YZ, Chu HC. The impact of IPACK combined with adductor canal block under ultrasound guidance on early motor function after total knee arthroplasty. Braz J Anesthesiol. 2022 Jan-Feb;72(1):110-114. doi: 10.1016/j.bjane.2021.04.012. Epub 2021 Apr 26. PMID 33915199
- [Background] Kim DH, Beathe JC, Lin Y, YaDeau JT, Maalouf DB, Goytizolo E, Garnett C, Ranawat AS, Su EP, Mayman DJ, Memtsoudis SG. Addition of Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee and Adductor Canal Block to Periarticular Injection Enhances Postoperative Pain Control in Total Knee Arthroplasty: A Randomized Controlled Trial. Anesth Analg. 2019 Aug;129(2):526-535. doi: 10.1213/ANE.0000000000003794. PMID 30234517
- [Background] Patterson ME, Vitter J, Bland K, Nossaman BD, Thomas LC, Chimento GF. The Effect of the IPACK Block on Pain After Primary TKA: A Double-Blinded, Prospective, Randomized Trial. J Arthroplasty. 2020 Jun;35(6S):S173-S177. doi: 10.1016/j.arth.2020.01.014. Epub 2020 Jan 15. PMID 32005622
- [Background] D'Souza RS, Langford BJ, Olsen DA, Johnson RL. Ultrasound-Guided Local Anesthetic Infiltration Between the Popliteal Artery and the Capsule of the Posterior Knee (IPACK) Block for Primary Total Knee Arthroplasty: A Systematic Review of Randomized Controlled Trials. Local Reg Anesth. 2021 May 12;14:85-98. doi: 10.2147/LRA.S303827. eCollection 2021. PMID 34012290